CLINICAL TRIAL: NCT05177276
Title: An Investigator Sponsored Phase I/II Study of Selinexor in Combination With Irinotecan in Adults With Solid Tumors
Brief Title: Selinexor Combination Ph 1 Study
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Martin Gutierrez (Other)
Collaborators: Hackensack Meridian Health (Other); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Martin Gutierrez, M.D.,Director Early Drug Development & Phase 1, Hackensack Meridian Health
Organization: Hackensack Meridian Health (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IST: PRO5126
Record Dates: First submitted 2019-06-17; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor Malignancy
MeSH Terms: interventions — selinexor; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose Level -1 (Experimental): Selinexor 12mg po twice weekly (Monday & Wednesday or Tuesday & Thursday); Irinotecan 50mg/m2 IV once daily on days 1, 8 & 15
  Interventions: Drug: Selinexor; Drug: Irinotecan
- Dose Level 1 (Experimental): Selinexor 15mg po twice weekly (Monday & Wednesday or Tuesday and Thursday); Irinotecan 75mg/m2 IV once daily on days 1, 8 & 15.
  Interventions: Drug: Selinexor; Drug: Irinotecan
- Dose Level 2 (Experimental): Selinexor 20mg po twice weekly (Monday & Wednesday or Tuesday and Thursday); Irinotecan 100mg/m2 IV once daily on days 1, 8 & 15.
  Interventions: Drug: Selinexor; Drug: Irinotecan
- Dose Level 3 (Experimental): Selinexor 30mg po twice weekly (Monday & Wednesday or Tuesday and Thursday); Irinotecan 75mg/m2 IV once daily on days 1, 8 & 15.
  Interventions: Drug: Selinexor; Drug: Irinotecan
- Dose Level 4 (Experimental): Selinexor 30mg po twice weekly (Monday & Wednesday or Tuesday and Thursday); Irinotecan 125mg/m2 IV once daily on days 1, 8 & 15.
  Interventions: Drug: Selinexor; Drug: Irinotecan

INTERVENTIONS:
Drug: Selinexor
  Other Names: KPT-330
Drug: Irinotecan
  Other Names: Camptosar

SUMMARY:
The purpose of this study is to determine the safety, tolerability and maximum tolerated dose of selinexor (KPT-330) in combination with Irinotecan in patients with solid tumors. A secondary purpose is to evaluate the pharmacokinetics (PK) of selinexor with irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed solid tumor malignancy that is metastatic or unresectable for which standard curative measures do not exist, or are associated with minimal patient survival benefit, and for whom irinotecan therapy may be appropriate.
* Any prior therapy must have been completed > 2 weeks prior to enrollment on the protocol in patients participating and must have recovered to eligibility levels (CTCAE grade </= 1) from prior toxicity. Prior radiation or surgery should have been completed > 2 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels.
* Age >/= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of selinexor in patients < 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase 1 combination trials.
* Eastern Cooperative Group (ECOG) performance status </= 2 (Karnofsky >/= 60%).
* Life expectancy >/= 3 months.
* Patients must have normal organ and marrow function as defined below:
* Absolute Neutrophil count >/= 1,500u/L
* Platelets >/= 125,000u/L
* Total Bilirubin </= 1.5x institution upper limit of normal
* AST (SGOT)/ALT(SGPT) </= 2.5x institutional upper limit of normal, if liver metastasis </= 5x institutional upper limit.
* Creatinine </= 1.5x institutional upper limit of normal. or
* Creatinine clearance >/= 50mL/minute for patients with creatininelevels > 1.5x institutional upper limit of normal.
* The effects of selinexor on the developing human fetus are unknown. For this reason, and because Irinotecan used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 30 days after completion of study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients who have previously

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or those who have not recovered from AEs due to agents administered more than 2 weeks earlier. Patients must be >/= 2 weeks since any investigational agent was administered as part of an exploratory IND study and should have recovered to eligibility levels from any toxicity.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrythmia, prolonged QTc interval (>500 msec), or psychiatric illness/social situations that would limit compliance with study requirements.
* In the Food and Drug Administration (FDA) Use-in-Pregnancy Ratings for Drugs, Irinotecan is classified as category D drugs, indicating that investigational or postmarketing data show risk to the fetus. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after completion of study. Should a woman become pregnant or suspect she is pregnant while participating in the study, she should inform her treating physician immediately. Because there is a risk for AEs in nursing infants secondary to treatment of the mother with these drugs, breastfeeding should be discontinued while the patient is on this trial and for 30 days after completion of treatment on this trial.
* Patients with known brain metastases are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status is stable with or without treatment without steroids (except for maintenance replacement doses of steroids).
* Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies or confirmed diagnosis of HIV infection, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are excluded from this trial.
* Grade >/= 3 toxicity related to irinotecan for patients who have received prior irinotecan.
* Both men and women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.03 | From date of first dose through study completion, an average of 1 year
  Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.03
Establish the maximum tolerated dose (MTD) for the combination of selinexor with Irinotecan. | From date of first dose through study completion, an average of 1 year
  Establish the maximum tolerated dose (MTD) for the combination of selinexor with Irinotecan.

CONTACTS AND LOCATIONS:
Locations (1):
- John Theurer Cancer Center at HackensackUMC, Hackensack, New Jersey, United States